CLINICAL TRIAL: NCT07145528
Title: Social Skills in Adult Patients Followed for Chronic Pain, Addiction, Intimate Partner Violence or Followed in Primary Care: A Comparative Observational Study
Brief Title: Social Skills in Chronic Pain, Addiction, Intimate Partner Violence and Primary Care
Acronym: Skills-PAVIP
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU Clermont-Ferrand; 2024-A00933-44 (Other: ANSM)
Record Dates: First submitted 2025-02-19; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-07

CONDITIONS: Social Skills; Primary Care
Keywords: intimate partner violence; addiction; chronic pain
MeSH Terms: conditions — Social Skills; Behavior, Addictive; Chronic Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Patients in Primary Care: A single E-case report form (CRF) for every group (a 45 minutes interview)
  Interventions: Other: Questionary with a case-report-form
- Patients with chronic pain: A single E-case report form (CRF) for every group (a 45 minutes interview)
  Interventions: Other: Questionary with a case-report-form
- Patients victims of violence: A single E-case report form (CRF) for every group (a 45 minutes interview)
  Interventions: Other: Questionary with a case-report-form
- Patients perpetrators of violence: A single E-case report form (CRF) for every group (a 45 minutes interview)
  Interventions: Other: Questionary with a case-report-form
- Patients with alcohol dependence: A single E-case report form (CRF) for every group (a 45 minutes interview)
  Interventions: Other: Questionary with a case-report-form

INTERVENTIONS:
Other: Questionary with a case-report-form — Questionary with : Gender, Age, Marital Status, medical history, Socio-économic description, skills assessment test written by R-Shankland, AUDIT-C, fargestrom, HAD, CAST, EPICE, Stroop-Test, Trail making test, Rosenberg Test

SUMMARY:
Context: psychosocial competencies (CPS) are higher cognitive functions defined by the ability to interact with others by adopting appropriate and positive behavior. They are defined among three axes: emotional skills, cognitive skills and social skills. Dysfunctions in social skills in adults are linked to substance use and abuse, sensitivity to pain, control of violence, and being a victim of violence. The links are bidirectional: both causes and consequences.

Objectives: Compare the level of psychosocial skills in patients presenting with a use disorder or chronic pain or being victims or perpetrators of domestic violence or patients followed in a primary care center without any of these histories, using the score obtained after passing a scale currently being validated in an adult population.

Secondary objectives Describe profiles of social skills dysfunction within each population Evaluate the link between alterations in CPS in the different populations and different sociodemographic, intrinsic or environmental criteria

Type of study: multicenter comparative cross-sectional study

Number of centers: twelve (6 multi-professional primary care health centers - 6 hospital centers)

Study description: Cross-sectional, multicenter study. The patients will be included consecutively over a one-year period at the time of their visit to the inclusion center.

Primary endpoint: score obtained for each of the 4 axes on the ad hoc psychosocial skills assessment test.

Number of subjects: 600 patients (60 in each group)

Inclusion criteria

* Patients aged 18 and over,
* Patients with chronic pain lasting at least 6 months,
* Patients with alcohol dependence,
* Patients victims of intra-family violence,
* Patients who commit intra-family violence,
* Patients followed in primary care and not presenting any of the 4 previous items,

Study procedure: each participant, regardless of population, will receive a single 45-minute interview consisting of a validated psychosocial skills assessment test, and a record of consumption status and medico-socio-economic history.

Data will be collected directly online, and the main analysis will be based on a comparative analysis of the level of social skills between the different groups for each of the four axes of the social skills assessment test.

DETAILED DESCRIPTION:
Context: psychosocial competencies (CPS) are higher cognitive functions defined by the ability to interact with others by adopting appropriate and positive behavior. They are defined among three axes: emotional skills, cognitive skills and social skills.

Social skills provide the conditions for modulating and controlling emotions, improving individual and social skills, making appropriate decisions, and resisting social conflicts. Poor social skills are linked to psychological disorders and psychiatric disorders such as mood disorders. Dysfunctions in social skills in adults are linked to substance use and abuse, sensitivity to pain, control of violence, and being a victim of violence. The links are bidirectional: both causes and consequences.

I

Objectives:

Main objective Compare the level of psychosocial skills in patients presenting with a use disorder or chronic pain or being victims or perpetrators of domestic violence or patients followed in a primary care center without any of these histories, using the score obtained after passing a scale currently being validated in an adult population,

Secondary objectives Describe profiles of social skills dysfunction within each population Evaluate the link between alterations in CPS in the different populations and different sociodemographic (gender, age, geographical area), intrinsic (executive functions) or environmental criteria (childhood trauma, precariousness...).

Type of study: multicenter comparative cross-sectional study

Number of centers: twelve (6 multi-professional primary care health centers - 6 hospital centers)

Study description: This is a cross-sectional, multicenter study in the RIPH 2 category. The patients will be included consecutively over a one-year period at the time of their visit to the emergency department. This is an interventional study in that a questionnaire will be administered, asking questions about sensitive data. There will be no follow-up.

Primary endpoint: score obtained for each of the four axes on the ad hoc psychosocial skills assessment test.

Number of subjects: 600 patients (60 in each group)

Inclusion criteria

* Patients aged 18 and over,
* Patients with chronic pain lasting at least 6 months,
* Patients with alcohol dependence,
* Patients victims of intra-family violence,
* Patients who commit intra-family violence,
* Patients followed in primary care and not presenting any of the 4 previous items,

Non inclusion criteria Patients not fluent in French, Patients with an unstabilized psychiatric disorder, Patients refusing to participate in the study. Persons not affiliated to a social security scheme or beneficiaries of a similar scheme, Subjects participating in another interventional research study with an exclusion period still in progress at the time of inclusion.

Patients deprived of liberty, under guardianship, curators or safeguard of justice.

Pregnant and breast-feeding women

Study procedure: each participant, regardless of population, will receive a single 45-minute interview consisting of a validated psychosocial skills assessment test, and a record of consumption status and medico-socio-economic history.

Data will be collected directly online, and the main analysis will be based on a comparative analysis of the level of social skills between the different groups for each of the four axes of the social skills assessment test.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18 and over Suicidal: Patients at risk of suicide, or Suicidal : Patients who have attempted suicide, or Primary care patients

Exclusion Criteria:

Patients not fluent in French, Patients with an unstabilized psychiatric disorder, Patients refusing to participate in the study. Persons not affiliated to a social security scheme or beneficiaries of a similar scheme, Pregnant and breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All eligible patients attending participating primary care centers during the study period
  All eligible patients consulting in the pain center of Clermont-Ferrand and Lyon, at the addiction center of Grenoble and Clermont-Ferrand, at the center for the care of perpetrators and victims of violence in Clermont-Ferrand during the study period
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Score of psychosocial skills | 5 minutes
  15-item scale, grouped into 4 axes: emotional (5 items), cognitive (4 items), social (4 items), assertiveness (2 items). The response modality is a Likert scale with 7 possible answers ranging from "Never" (1) to "Always" (7). The alpha-cronbach coefficient was 0.754 for the cognitive axis, 0.731 for the social axis and 0.654 for the emotional axis

SECONDARY OUTCOMES:
Results of the others test | 45 minutes
  Sociodemographics criterias, intrinsics criteria, medical history, patient's health

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Laporte, Pr, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No